CLINICAL TRIAL: NCT02165995
Title: Use of Navigated Transcranial Magnetic Stimulation (nTMS) in Generated Motor and Language Mapping to Evaluate Brain Recovery and Plasticity Following Brain Tumor Surgery in or Adjacent to Eloquent Cortex
Brief Title: Use of Navigated Transcranial Magnetic Stimulation (nTMS) in Generated Motor and Language Mapping to Evaluate Brain Recovery Following Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0711; NCI-2015-01905 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-06-11; First posted 2014-06-18 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Brain Tumor
Keywords: Brain Tumor; Glioma; Tumor resection; Navigated Transcranial Magnetic Stimulation; nTMS; Brain mapping; Motor function; Speech function; Speech mapping
MeSH Terms: conditions — Brain Neoplasms; Glioma; Speech

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Navigated Transcranial Magnetic Stimulation (nTMS) (Experimental): Participant assessed by nTMS system before surgery, then again at 1, 3, 6, and 12 months following surgery. Motor mapping and speech mapping performed at these visits. This should take about 1½-2 hours to complete.
  Interventions: Procedure: Motor Mapping; Procedure: Speech Mapping

INTERVENTIONS:
Procedure: Motor Mapping — Motor mapping performed using nTMS system before surgery, then again at 1, 3, 6, and 12 months following surgery. Pads to monitor movements placed on face, arms and legs. A coil that is used to deliver stimulation will be placed on head. During stimulation, participant be asked to move certain muscles and will be monitored for motor responses over the course of 20 to 30 minutes.
Procedure: Speech Mapping — Speech mapping performed using nTMS system before surgery, then again at 1, 3, 6, and 12 months following surgery. Participant shown 95 black-and-white drawings of common objects and asked to name them. During stimulation, participant asked to name the objects again and will be monitored for changes in speech or delays. This should take about 1½-2 hours to complete.

SUMMARY:
The goal of this clinical research study is to learn about using Navigated Transcranial Magnetic Stimulation (nTMS) in patients having surgery to remove a brain tumor in areas of the brain that control movement (motor function) and/or speech.

nTMS is a system designed to map the brain's function relating to movement and speech.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will be assessed by the nTMS system before surgery and then at the same time as your routine follow-up visits, about 1, 3, 6, and 12 months after surgery.

At each visit, the following will occur:

* For motor mapping, pads to monitor your movements will be placed on your face, arms and legs. A coil that is used to deliver stimulation will be placed on your head. During stimulation, you will be asked to move certain muscles and will be monitored for motor responses over the course of 20 to 30 minutes. You may feel a mild tingling sensation in your arms and/or legs during stimulation.
* For speech mapping, you will be shown 95 black-and-white drawings of common objects and asked to name them. During stimulation, you will be asked to name the objects again and will be monitored for changes in speech or delays. You may feel a mild tingling sensation and contraction of the muscles in the face during stimulation. This should take about 1½-2 hours to complete.

You will sign a separate consent form that describes the surgery you will have and its risks in more detail. Information collected during surgery will be compared to nTMS information collected before and after surgery.

Your nTMS data, health information from your routine physical exams, and data about your motor and speech function collected during surgery will be analyzed by researchers. Basic information (such as your age, sex, and race) will also be collected from your medical record.

Length of Study:

Your participation in this study will be over after your last (12-month) study visit.

This is an investigational study. The nTMS system is FDA approved to map the brain's function relating to movement and speech. Using the nTMS system before and after surgery to check movement and speech function in patients with brain tumors in these areas is investigational.

Up to 20 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a new or recurrent, presumed or documented, diagnosis of primary or secondary brain tumor in or adjacent to eloquent brain areas (motor, SMA and language) who are scheduled to undergo tumor resection.
2. Patients must sign an informed consent.

Exclusion Criteria:

1. Patients with a history of uncontrolled seizures
2. Patients with metal implant or a cardiac pacemaker

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Pre and Post-Operative Functional Outcomes Using Navigated Transcranial Magnetic Stimulation (nTMS) | 12 months
  Data obtained using nTMS correlated with data collected intraoperatively during direct electrical stimulation (DES). nTMS stimulation also correlated with neurological status and functional recovery after surgery. The Chi-square or Fisher's exact tests used to explore associations between categorical variables. T-tests, Wilcoxon rank sum tests, or regression models used for continuous variables.

CONTACTS AND LOCATIONS:
Overall Officials: Sujit Prabhu, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org